CLINICAL TRIAL: NCT04887415
Title: Safety, Feasibility, and Impact of Preoperative Respiratory Strength Training in Cardiac Surgical Patients
Brief Title: Respiratory Strength Training in Cardiac Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Speech-Language-Hearing Foundation (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB202100993; OCR40654 (Other: UF OnCore)
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Thoracic Diseases; Surgery; Surgery--Complications; Dysphagia
MeSH Terms: conditions — Cardiovascular Diseases; Thoracic Diseases; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Longitudinal pilot cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enrolled Participants (Experimental): Enrolled cardiac surgical patients who underwent a 4 weeks of preoperative respiratory strength training (RST) program using two respiratory strength training devices.
  Interventions: Behavioral: Respiratory Strength Training (RST) Program

INTERVENTIONS:
Behavioral: Respiratory Strength Training (RST) Program — Participants will complete RST exercises 5 days per week by performing 5 sets of 5 repetitions of both expiratory and inspiratory muscle strength training (a total of 50 repetitions per day). Trainer devices will be calibrated to 50% of participants' maximum expiratory pressure (MEP) and maximum inspiratory pressure (MIP) as determined via respiratory assessment prior to and during the RST program.

SUMMARY:
Swallowing difficulty (dysphagia) is a common postoperative complication in patients who undergo cardiac surgical procedures. Postoperative dysphagia in cardiac surgical patients is associated with negative health-related outcomes including increased rates of pneumonia, reintubation, and death as well as increased length of hospital stay and costs of care. This study will examine the safety, feasibility, and impact of preoperative respiratory strength training (RST) on swallowing and associated health-related outcomes in cardiac surgical patients. We hypothesize that preoperative RST will be safe, well-tolerated, and lead to improved swallowing and health-related outcomes in cardiac surgical patients.

DETAILED DESCRIPTION:
Enrolled research participants will undergo baseline assessments of pulmonary function: maximum expiratory pressure (MEP), maximum inspiratory pressure (MIP), cough function (voluntary PEF and cough spirometry), and will complete self-reported dyspnea using the validated London Chest Activity of Daily Living (LCADL) scale. Following baseline testing, participants will complete a respiratory strength training program (RST) in the home via telehealth with one in-person home therapy session conducted at each participant's midpoint to reassess MEP and MIP and to recalibrate the respiratory strength trainer devices. After the prescribed RST program, participants will complete a second post-RST preoperative assessment. All pulmonary function measures will be performed by a research SLP in accordance with standardized protocols and guidelines from the American Thoracic Society 12-14 with research participants in an upright seated position with nose clips in place. A swallowing examination (FEES) will be completed both pre and post surgery to assess any impact on swallowing safety.

Respiratory Assessment:

MEP and MIP measurements will be obtained using a MicroRPM handheld menometry device (MicroDirect). For MEP testing, research participants will be instructed to take a deep breath in, place their mouth around the mouthpiece, and blow out as forcefully as possible. As needed, the research SLP will assist with lip seal by holding the sides of participant's cheeks to prevent air leakage. For MIP testing, research participants will be instructed to expel all the air out of their lungs, place their mouth around the mouthpiece, and breathe in as forcefully as possible. Each participant will perform 3 MEP and MIP trials. Average MEP and MIP values will be used to calibrate expiratory and inspiratory devices and for subsequent analyses.

Respiratory Strength Training (RST) Program:

The RST program consists of expiratory muscle strength training (EMST) and inspiratory muscle strength training (IMST) using the EMST-75 Lite or the EMST-150 and the IA-150 devices (Aspire Products), respectively. Trainer devices will be calibrated to a 50% load of individualized MEP and MIP values. The CS patients will perform 25 repetitions each (5 sets of 5 repetitions) of the expiratory and inspiratory exercises, 5 days/week leading up to their surgical procedure. The patients will be given training logs to track completion of the RST exercises to measure adherence.

Telehealth sessions:

Telehealth sessions will be conducted by a research speech-language pathologist (SLP) at least once per week via a secure version of Zoom. During telehealth sessions, the research SLP will ensure that participants performed the prescribed exercises with correct form, completed a safety and adverse event check, answered participant questions, assisted with adherence issues, monitored adverse events, and aided participants in adjusting the resistance of the expiratory and inspiratory training devices based on participant exertion ratings using the Borg Category Ratio 10 Scale.11 During the adverse event check, the research SLP will ask research participants if they were experiencing any pain, fatigue, discomfort, or other adverse events related to the RST protocol. Attendance for telehealth sessions will be tracked.

Home Visits:

In addition to weekly telehealth sessions, a home visit will be conducted by a research SLP midway through the RST program. During the home visit, the research SLP will perform check-ins similar to telehealth sessions, retest MEP and MIP, and recalibrate the training devices to meet the 50% training load target.

Fiberoptic Endoscopic Evaluation of Swallowing (FEES):

Participants will undergo a FEES exam in a dedicated room in the preoperative clinic or the ARC lab before and after completing the RST program using an Olympus flexible video HD Rhino Laryngoscope connected to a portable video processor and light source. To ensure patient comfort, a water-soluble lubricant and, per participant preference, a topical numbing-agent (i.e., lidocaine) will be applied to the naris, and the laryngoscope will be passed trans-nasally through the nasopharynx and hypopharynx until an optimal position is obtained. A standardized FEES protocol will be used that includes a combination of voicing and swallowing tasks. At the completion of the swallowing trials, the laryngoscope will be carefully removed. Blinded analysis of the swallowing exam will be performed.

Statistical Analysis:

Demographic information and pulmonary and cough function data will be exported directly from our secure online database, REDCap, into JMP version 16.1.020 and Prism version 9.4.1 (GraphPad Software) for statistical analyses. Descriptive statistics will be used to summarize demographic information and pulmonary and cough function data. Intraclass correlation coefficients (ICCs) with 95%confidence intervals (CI) will be used to calculate inter-rater and intrarater reliability for voluntary cough spirometry metrics. Mean differences with 95% CIs will be calculated, and the Wilcoxon signed-rank test will be performed to assess pre-RST to post-RST changes in pulmonary and cough function.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18-90 years old.
2. Not pregnant.
3. Undergoing planned cardiac surgery via sternotomy &/or extended thoracotomy & seen in the UF Health preoperative clinic.
4. Confirmed COVID-19 negative test and/or no recent COVID-19 symptoms
5. Has access to a computer, tablet, or electronic device with a stable internet connection for telehealth sessions.
6. Willing to undergo testing procedures and complete the exercise training program

Exclusion Criteria:

1. Individuals under the age of 18 or over the age of 90.
2. Pregnant women.
3. Positive for COVID-19 or symptoms of COVID-19
4. No access to a computer, tablet, or electronic device &/ a stable internet connection for telehealth sessions.
5. Unwilling to undergo testing procedures and/or complete the exercise training program.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, Ph.D., Principal Investigator — University of Florida
Locations (1):
- Cardiovascular Clinic and Thoracic/Cardiovascular Surgery at UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enrolled Participants
Started | 25
Completed | 23
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Surgery Type [Count of Participants; unit: Participants]
  Mitral Valve | 8
  Aorta Graft | 3
  Aortic Arch | 3
  Maze Procedure | 3
  Multiple Valve Replacement | 2
  Aortic Root | 1
  CABG | 1
  LVAD | 1
  Tricuspid Valve | 1
  Mini Aortic Valve | 1
  Atrial Appendage Ligation with an Atriclip | 1

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Respiratory Strength Training
Description: Number of respiratory strength training repetitions
Time Frame: 4 weeks
Measure: Count of Units; unit: Repetitions
Units Other Than Participants: Repetitions
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 23
Number analyzed (Repetitions) | 36650
Repetitions | 35750

2. Primary Outcome: Attendance at Telehealth Sessions
Description: Number of Telehealth sessions completed
Time Frame: 4 weeks
Measure: Count of Units; unit: Telehealth Sessions
Units Other Than Participants: Telehealth Sessions
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 23
Number analyzed (Telehealth Sessions) | 135
Telehealth Sessions | 135

3. Primary Outcome: Change in Maximum Expiratory Pressure (MEP) Between Pre and Post Respiratory Strength Training
Description: A measure of maximum expiratory respiratory strength (in cmH2O) prior to and after completing RST program.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 23
cmH2O
  Pre-RST | 105.6 (40.9)
  Post-RST | 120.9 (49.7)

4. Primary Outcome: Change in Maximum Inspiratory Pressure (MIP) Pre and Post Respiratory Strength Training
Description: A measure of maximum inspiratory strength (in cmH2O) prior to and after completing RST program.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 23
cmH2O
  Pre-RST | 73.2 (26.4)
  Post-RST | 88.1 (30.9)

5. Primary Outcome: Change in Cough Peak Expiratory Flow Between Pre and Post Respiratory Strength Training
Description: A measure of cough strength (in L/min of air flow) prior to and after completing RST program.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 23
L/min
  Pre-RST | 337.7 (128.5)
  Post-RST | 352.7 (144.3)

6. Primary Outcome: Change in Worst Penetration-aspiration Scale (PAS) Score From Pre and Post Surgical Fiberoptic Endoscopic Evaluation of Swallowing (FEES).
Description: The Penetration-Aspiration Scale (PAS) is a validated 8-point ordinal rating scale that measures the depth of airway invasion of bolus material and patient response during swallowing. PAS scores range from 1 to 8, with a score of 1 indicating a safe swallow (no penetration or aspiration of bolus material) (best score) and 8 indicating silent aspiration (bolus material reached below the level of the vocal folds and no response / effort to eject material was made) (worst score). After analysis of the FEES examination, the worst overall PAS score across was determined across all bolus types administered during the exam and recorded for both the preoperative FEES exam and the post-operative FEES exam.
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Participants - Preoperative PAS Outcomes: Enrolled cardiac surgical patients who underwent a 4 weeks of preoperative respiratory strength training (RST) program using two respiratory strength training devices.
  A fiberoptic endoscopic evaluation of swallowing (FEES) was performed after RST training, prior to their scheduled cardiac surgery. Analysis of the FEES procedure included evaluation of the worst overall PAS score during the FEES examination.
- Enrolled Participants - Post-Operative PAS Outcomes: Enrolled cardiac surgical patients who underwent a 4 weeks of preoperative respiratory strength training (RST) program using two respiratory strength training devices.
  A fiberoptic endoscopic evaluation of swallowing (FEES) was performed after their scheduled cardiac surgery. Analysis of the FEES procedure included evaluation of the worst overall PAS score during the FEES examination.
Arm/Group | Enrolled Participants - Preoperative PAS Outcomes | Enrolled Participants - Post-Operative PAS Outcomes
Number analyzed (Participants) | 23 | 22
Participants
  Worst PAS Score = 1 | 13 | 2
  Worst PAS Score = 2 | 1 | 0
  Worst PAS Score = 3 | 4 | 9
  Worst PAS Score = 4 | 2 | 0
  Worst PAS Score = 5 | 1 | 4
  Worst PAS Score = 6 | 0 | 1
  Worst PAS Score = 7 | 0 | 1
  Worst PAS Score = 8 | 2 | 5

ADVERSE EVENTS:
Time Frame: From participant enrollment date through study completion (participant is discharged from hospital following cardiac surgery), an average of 8 weeks.
Arm/Group | Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 8/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Participants (N=25)
Pain (mild) (General disorders) | 2 (25)
Dizziness (General disorders) | 7 (25)
Migraine (General disorders) | 1 (25)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 (25)
Bloody Nose (Respiratory, thoracic and mediastinal disorders) | 1 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT04887415/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04887415/ICF_001.pdf